CLINICAL TRIAL: NCT02328508
Title: Hyperbaric Oxygen Therapy in Diabetics With Chronic Foot Ulcers and Improvement of Quality of Life
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chen-Yu Chen (Other)
Collaborators: I-Shou University (Other)
Responsible Party: Sponsor-Investigator, Chen-Yu Chen, Registered Nurse, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-0876B, 101-0507C
Record Dates: First submitted 2014-12-25; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Diabetic Foot Ulcer; Diabetes
Keywords: hyperbaric oxygen therapy; diabetic foot ulcer; wound healing; inflammation; glycemic control; amputation; bacterial infection; quality of life
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Inflammation; Bacterial Infections | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hyperbaric oxygen therapy (Experimental): The experimental group received treatments in a hyperbaric chamber for 120-min per session, once per day, and five days per week for four consecutive weeks (20 treatment sessions).
  Interventions: Device: Hyperbaric oxygen therapy
- Control (No Intervention): The control group received only routine care.

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — HBOT was carried out in a hyperbaric chamber for 120-min per session, five days a week for four consecutive weeks (20 treatment sessions).
  Other Names: HBOT
  Arms: hyperbaric oxygen therapy

SUMMARY:
This study evaluated the effect of hyperbaric oxygen therapy (HBOT) on wound healing, inflammation index, glycemic control, amputation rate, survival rate of tissue, bacterial wound cultures, and quality of life (QOL) in diabetic foot ulcer (DFU) patients with diabetes.

DETAILED DESCRIPTION:
OBJECTIVE - This study evaluated the effect of hyperbaric oxygen therapy (HBOT) on wound healing, inflammation index, glycemic control, amputation rate, survival rate of tissue, bacterial wound cultures, and quality of life (QOL) in diabetic foot ulcer (DFU) patients with diabetes.

RESEARCH DESIGN AND METHODS - This study was a randomized, single-center clinical trial. The effects of HBOT on patients in the experimental group were compared with the control group received only routine care. HBOT was carried out in a hyperbaric chamber for 120-min per session, five days a week for four consecutive weeks (20 treatment sessions). Data were collected at 4 segments: pre-treatment (before first administration of HBOT; T1), during treatment (at the tenth administration of HBOT; T2), post-treatment (at the twentieth administration of HBOT; T3), and treatment follow-up (two weeks after the last therapy ended; T4).

ELIGIBILITY:
Inclusion Criteria:

* over 20 years of age
* a history of diabetes and a diagnosis of diabetic foot
* a wound classification of Grade 3 or below
* clear conscious and willing to participate in this study
* a signed consent form

Exclusion Criteria:

* less than 20 years of age, unwilling to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
wound healing | 4 weeks
  The Wagner Ulcer Grade Classification System for wound physiological index

SECONDARY OUTCOMES:
inflammation index | 4 weeks
  Erythrocyte sedimentation rate, ESR; C-reactive protein, CRP
amputation rate | 4 weeks
  Number of patients undergo surgical removal of a limb
survival rate of tissue in the affected limb | 4 weeks
  blood flow perfusion scan
bacteriological wound cultures | 4 weeks
  collect and culture bacteria from the wound to see whether a wound is infected, to identify the bacteria causing the infection
glycemic control | 4 weeks
  Glycated Hemoglobin, HbA1c Hemoglobin, HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Yu Chen, Master, Principal Investigator — Chang Gung Memorial Hospital